CLINICAL TRIAL: NCT02819089
Title: Recovery Profiles After c Spine Surgery: With or Without Dexmedetomidine as an Anesthetic Adjuvant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 018/2559(EC1)
Record Dates: First submitted 2016-06-15; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Cervical Spondylosis
Keywords: anterior cervical spine surgery; ACDF; Dexmedetomidine; Anesthesia; Agitation; Riker sedation agitation scores
MeSH Terms: conditions — Spondylosis; Psychomotor Agitation | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Active Comparator): Demedetomidine infusion (2mcg/ml); loading 0.5 mcg/kg for 30 min (BW/2 ml/h for 30 min), then 0.5 mcg/kg (BW/4 ml/h) until 30 minutes before finish the operation.
  Interventions: Drug: Dexmedetomidine
- NSS (Placebo Comparator): NSS loading BW/2 ml/h for 30 min, then BW/4 ml/h until 30 minutes before finish the operation.
  Interventions: Other: NSS

INTERVENTIONS:
Drug: Dexmedetomidine — Demedetomidine infusion (2mcg/ml); loading 0.5 mcg/kg for 30 min (BW/2 ml/h for 30 min), then 0.5 mcg/kg (BW/4 ml/h) until 30 minutes before finish the operation.
  Other Names: Precedex
  Arms: Dexmedetomidine
Other: NSS — NSS infusion; loading BW/2 ml/h for 30 min, then BW/4 ml/h until 30 minutes before finish the operation.
  Other Names: Narmal saline, 0.9%NaCl
  Arms: NSS

SUMMARY:
The purpose of this study is to determine the recovery profiles after general anesthesia in patient undergoing anterior cervical spine surgery. This study will compare the Riker sedation agitation scores between two groups, with or without dexmedetomidine as an anesthetic adjuvant.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* elective case for ACDF surgery
* plan for extubation after surgery

Exclusion Criteria:

* SBP>140 mmHg
* CAD
* HR<50 BPM, heart block
* motor weakness > grade 4
* BMI >30
* allergic to dexmedetomidine, fentanyl

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Riker sedation agitation scores | before extubation
  After finish the operation, Desflurane will be stopped. All patients will be received the neuromuscular reversal drugs and TOF ratio > 0.9. All patients will be evaluated by Riker sedation agitation score before extubation and re-evaluated again at 15 minutes after extubation.
  Riker sedation agitation scores
  1. Dangerous agitation: trying to get out of bed, pulling out tube, thrashing
  2. Very agitated: may require physical restraint, unable to calm with verbal instructions.
  3. Agitated: mild agitation and anxiety but calm down with verbal instructions.
  4. Calm and cooperative: aroused easily and follows commands
  5. Sedated: difficult to aroused, but does arouse to verbal or physical stimuli, able to follow simple commands
  6. Very sedated: does not follow commands but arouses to physical stimulation
  7. Unarousable: little or no response to noxious stimuli

SECONDARY OUTCOMES:
Fentanyl consumption | during surgery
  After finish the operation, the total of fentanyl consumption during the operation will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Busara Sirivanasandha, MD, Principal Investigator — Department of Anesthesiology, Siriraj Hospital, Mahidol University
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lepouse C, Lautner CA, Liu L, Gomis P, Leon A. Emergence delirium in adults in the post-anaesthesia care unit. Br J Anaesth. 2006 Jun;96(6):747-53. doi: 10.1093/bja/ael094. Epub 2006 May 2. PMID 16670111
- [Background] Yu D, Chai W, Sun X, Yao L. Emergence agitation in adults: risk factors in 2,000 patients. Can J Anaesth. 2010 Sep;57(9):843-8. doi: 10.1007/s12630-010-9338-9. Epub 2010 Jun 5. PMID 20526708
- [Background] Khan ZP, Ferguson CN, Jones RM. alpha-2 and imidazoline receptor agonists. Their pharmacology and therapeutic role. Anaesthesia. 1999 Feb;54(2):146-65. doi: 10.1046/j.1365-2044.1999.00659.x. PMID 10215710
- [Background] Maze M, Scarfini C, Cavaliere F. New agents for sedation in the intensive care unit. Crit Care Clin. 2001 Oct;17(4):881-97. doi: 10.1016/s0749-0704(05)70185-8. PMID 11762266
- [Background] Kim HS, Byon HJ, Kim JE, Park YH, Lee JH, Kim JT. Appropriate dose of dexmedetomidine for the prevention of emergence agitation after desflurane anesthesia for tonsillectomy or adenoidectomy in children: up and down sequential allocation. BMC Anesthesiol. 2015 May 27;15:79. doi: 10.1186/s12871-015-0059-z. PMID 26012345
- [Background] Polat R, Peker K, Baran I, Bumin Aydin G, Topcu Guloksuz C, Donmez A. Comparison between dexmedetomidine and remifentanil infusion in emergence agitation during recovery after nasal surgery: A randomized double-blind trial. Anaesthesist. 2015 Oct;64(10):740-6. doi: 10.1007/s00101-015-0077-8. Epub 2015 Sep 2. PMID 26329913
- [Background] Gopalakrishna KN, Dash PK, Chatterjee N, Easwer HV, Ganesamoorthi A. Dexmedetomidine as an Anesthetic Adjuvant in Patients Undergoing Transsphenoidal Resection of Pituitary Tumor. J Neurosurg Anesthesiol. 2015 Jul;27(3):209-15. doi: 10.1097/ANA.0000000000000144. PMID 25493927
- [Background] Anjum N, Tabish H, Debdas S, Bani HP, Rajat C, Anjana Basu GD. Effects of dexmedetomidine and clonidine as propofol adjuvants on intra-operative hemodynamics and recovery profiles in patients undergoing laparoscopic cholecystectomy: A prospective randomized comparative study. Avicenna J Med. 2015 Jul-Sep;5(3):67-73. doi: 10.4103/2231-0770.160231. PMID 26229757
- [Background] Mariappan R, Ashokkumar H, Kuppuswamy B. Comparing the effects of oral clonidine premedication with intraoperative dexmedetomidine infusion on anesthetic requirement and recovery from anesthesia in patients undergoing major spine surgery. J Neurosurg Anesthesiol. 2014 Jul;26(3):192-7. doi: 10.1097/ANA.0b013e3182a2166f. PMID 23887684
- [Background] Ge DJ, Qi B, Tang G, Li JY. Intraoperative Dexmedetomidine Promotes Postoperative Analgesia in Patients After Abdominal Colectomy: A Consort-Prospective, Randomized, Controlled Clinical Trial. Medicine (Baltimore). 2015 Sep;94(37):e1514. doi: 10.1097/MD.0000000000001514. PMID 26376397
- [Background] Anastasian ZH, Gaudet JG, Levitt LC, Mergeche JL, Heyer EJ, Berman MF. Factors that correlate with the decision to delay extubation after multilevel prone spine surgery. J Neurosurg Anesthesiol. 2014 Apr;26(2):167-71. doi: 10.1097/ANA.0000000000000028. PMID 24296539
- [Background] Cavallone LF, Vannucci A. Review article: Extubation of the difficult airway and extubation failure. Anesth Analg. 2013 Feb;116(2):368-83. doi: 10.1213/ANE.0b013e31827ab572. Epub 2013 Jan 9. PMID 23302983
- [Background] Karwacki Z, Niewiadomski S, Rzaska M, Witkowska M. The effect of bispectral index monitoring on anaesthetic requirements in target-controlled infusion for lumbar microdiscectomy. Anaesthesiol Intensive Ther. 2014 Sep-Oct;46(4):284-8. doi: 10.5603/AIT.2014.0046. PMID 25293480
- [Background] Tsai CJ, Chu KS, Chen TI, Lu DV, Wang HM, Lu IC. A comparison of the effectiveness of dexmedetomidine versus propofol target-controlled infusion for sedation during fibreoptic nasotracheal intubation. Anaesthesia. 2010 Mar;65(3):254-9. doi: 10.1111/j.1365-2044.2009.06226.x. Epub 2010 Jan 22. PMID 20105150
- [Background] Terao Y, Ichinomiya T, Higashijima U, Tanise T, Miura K, Fukusaki M, Sumikawa K. Comparison between propofol and dexmedetomidine in postoperative sedation after extensive cervical spine surgery. J Anesth. 2012 Apr;26(2):179-86. doi: 10.1007/s00540-011-1300-7. Epub 2011 Dec 16. PMID 22173570
- [Background] Ge DJ, Qi B, Tang G, Li JY. Intraoperative Dexmedetomidine Promotes Postoperative Analgesia and Recovery in Patients after Abdominal Colectomy: A CONSORT-Prospective, Randomized, Controlled Clinical Trial. Medicine (Baltimore). 2015 Oct;94(43):e1727. doi: 10.1097/MD.0000000000001727. PMID 26512563